CLINICAL TRIAL: NCT03243136
Title: The Association Between Food Insecurity and Incident Type 2 Diabetes in Canada: A Population-based Cohort Study
Status: Completed | Type: Observational
Sponsor: Christopher Tait (Other)
Collaborators: Ontario Agency for Health Protection and Promotion (Other Government)
Responsible Party: Sponsor-Investigator, Christopher Tait, PhD Candidate, University of Toronto
Organization: University of Toronto (Other)
Other Study IDs: PROTOCOL REFERENCE # 32143
Record Dates: First submitted 2017-08-04; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exposure of interest is food insecurity — Households were considered food insecure if any of the following conditions were met in the past 12 months: 1) a member of the household worried that there would not be enough food to eat because of a lack of money, 2) a member's food intake was reduced as a result of there not being enough food to eat, or 3) the desired variety or quality of foods was not eaten because of a lack of money. This exposure variable was operationalized as a binary variable with levels of food secure vs. food insecure.

SUMMARY:
A pervasive and persistent finding is the health disadvantage experienced by those in food insecure households. While clear associations have been identified between food insecurity and diabetes risk factors, less is known about the relationship between food insecurity and incident type 2 diabetes.

The objective of this study is to investigate the association between household food insecurity and the future development of type 2 diabetes.

The investigators used data from Ontario adult respondents to the 2004 Canadian Community Health Survey, linked to health administrative data (n = 4,739). Food insecurity was assessed with the Household Food Security Survey Module and incident type 2 diabetes cases were identified by the Ontario Diabetes Database. Multivariable adjusted Cox proportional hazards models were used to estimate hazard ratios (HRs) and 95% confidence intervals (CIs) for type 2 diabetes as a function of food insecurity.

DETAILED DESCRIPTION:
Globally, there are over 200 million people living with type 2 diabetes. Aging populations, steadily increasing obesity rates, increases in sedentary behaviours, and decreases in diabetes-related mortality signal that the global prevalence of type 2 diabetes will continue to grow.

In Canada, type 2 diabetes is one of the most prevalent chronic conditions and is the 7th leading cause of mortality. Over the last decade, the prevalence of type 2 diabetes in Canada has increased by 72%, with 11 million Canadians currently living with diabetes or pre-diabetes. This number is expected to rise to 13.9 million (33% of Canadians) by 2026.

Much of the body of literature concerning type 2 diabetes focuses on management and control. Research that is geared towards prevention focuses heavily on the modification of individual risk behaviours, while less attention is given to the broader social determinants of increased type 2 diabetes risk.

Household food security is a broad measure of socioeconomic status that is not traditionally included in health research. Household food insecurity is experienced when there is uncertainty regarding, or disruption in, food intake or eating patterns by at least one member of a household due to financial constraints, resulting in inadequate or insecure access to food.

Food insecurity has been identified as a significant social and health problem in Canada . It was first measured in 2004, where it was estimated that 9.2% of Canadian households were food insecure. The most recent estimate from 2014 indicates that this number has risen to 12%, representing 3.2 million Canadians.

While there exists the perception that food insecurity leads to caloric restriction, food insecurity has been associated with lower nutrient intakes and consumption of a less healthy diet compared to those who are food secure. Prior evidence from cross-sectional studies has demonstrated that there is an association between food insecurity and chronic disease risk including hypertension, cardiovascular disease, and type 2 diabetes.

Though clear associations have been identified between food insecurity and diabetes risk factors such as dietary consumption, weight gain, and obesity, less is known about the direct relationship between food insecurity and incident type 2 diabetes. Moreover, limited studies have investigated this association longitudinally in a population-based sample.

Prospective, longitudinal assessment is critical as cross-sectional studies lack the ability to infer the direction of the relationship between food insecurity and type 2 diabetes. For example, the 'health selection' hypothesis has been studied, positing that a decline in health status may precede and ultimately cause downward social mobility and a decrease in income leading to food insecurity. Consequently, this theory presents evidence for reverse causation, by which poor health may precede financial difficulties, especially in cases where early age of diagnosis, and thus longer duration of disease, might predispose individuals to being in a food insecure household.

Current estimates of the future health consequences associated with food insecurity are needed to inform health decision-makers of potential areas for upstream intervention to alleviate the burden type 2 diabetes places on the Canadian healthcare system. Data linkages provide a novel opportunity to study this relationship in a prospective, population-based sample. Accordingly, the objectives of this study are to estimate the risk of type 2 diabetes as a function of food insecurity in the Canadian population, and to investigate the extent to which this association may be mediated by obesity.

ELIGIBILITY:
The investigators restricted the analyses to individuals ≥ 18 years of age at baseline who were successfully linked to the Ontario Diabetes Database (n = 5,539). The investigators further excluded pregnant women from the sample to increase the accuracy of body weight measurements (n = 36), prevalent cases of diabetes before respondents' 2004 Canadian Community Health Survey interview date (n = 636), underweight individuals (n = 112), and those who had missing information on food security status (n = 16). After these exclusions, the analytic cohort consists of 4,739 individuals, 2,050 men and 2,689 women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators used data from Ontario adult respondents to Cycle 2.2 of Canadian Community Health Survey conducted in 2004, deterministically linked to the Ontario Diabetes Database. The Canadian Community Health Survey is a cross-sectional survey administered by Statistics Canada that uses a multi-stage, stratified, clustered probability sample that is representative of 98% of the Canadian population. Those who are full-time members of the Canadian Forces, reside on First Nations Reserves or Crown Lands, are institutionalized, and who reside in certain remote areas reflect the 2% of the population not captured by the survey. Detailed descriptions of the survey methodology have been published elsewhere.
Sampling Method: Probability Sample
Enrollment: 4739 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Type 2 diabetes | 2004-2016
  Incident type 2 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Tait, PhD(c), Principal Investigator — University of Toronto - Dalla Lana School of Public Health

IPD SHARING:
Plan to Share IPD: No